CLINICAL TRIAL: NCT06134804
Title: A Phase 3 Randomized Double-blind Controlled Study to Evaluate the Immunogenicity, Safety, and Reactogenicity of ExPEC9V and High-dose Quadrivalent Influenza Vaccine, With and Without Co-administration, in Adults Aged 65 Years or Older
Brief Title: A Study of 9-valent Extraintestinal Pathogenic Escherichia Coli Vaccine (ExPEC9V) and High-dose Quadrivalent Influenza Vaccine, With and Without Co-administration, in Adults Aged 65 Years or Older
Acronym: Engage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR109338; 2023-504168-40-00 (Registry Identifier: EUCT number); VAC52416BAC3002 (Other: Janssen Research & Development LLC)
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Invasive Extraintestinal Pathogenic Escherichia Coli Disease (IED) Prevention

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Coadministration (CoAd) Group (Experimental): Participants will receive intramuscular (IM) injection of 9-valent extraintestinal pathogenic Escherichia coli vaccine (ExPEC9V) along with high-dose (HD) quadrivalent influenza vaccine, concomitantly, on Day 1 and placebo on Day 30.
  Interventions: Biological: ExPEC9V; Biological: Placebo; Biological: HD quadrivalent influenza vaccine
- Group 2: Control Group (Experimental): Participants will receive IM injection of matching placebo along with HD quadrivalent influenza vaccine, concomitantly, on Day 1 and ExPEC9V on Day 30.
  Interventions: Biological: ExPEC9V; Biological: Placebo; Biological: HD quadrivalent influenza vaccine

INTERVENTIONS:
Biological: ExPEC9V — ExPEC9V will be administered as an IM injection.
  Other Names: VAC52416; JNJ-78901563
Biological: Placebo — Placebo will be administered as an IM injection.
Biological: HD quadrivalent influenza vaccine — HD quadrivalent influenza vaccine will be administered as IM injection.

SUMMARY:
The purpose of this study is to show that high-dose quadrivalent seasonal influenza vaccine (HD QIV) given together with 9-valent extraintestinal pathogenic Escherichia coli vaccine (ExPEC9V) does not induce lower antibody response against each of the 4 influenza vaccine strains, as compared to HD QIV given alone and further show that ExPEC9V given together with HD QIV does not induce lower antibody response against each of the vaccine O-serotype antigens, as compared to ExPEC9V given alone.

ELIGIBILITY:
Inclusion Criteria:

* Must be medically stable at the time of vaccination such that, according to the judgment of the investigator, hospitalization within the study period is not anticipated and the participant appears likely to be able to remain on study through the end of protocol specified follow-up. A stable medical condition is defined as disease not requiring significant change in therapy during the 6 weeks before enrollment and when hospitalization for worsening of the disease is not anticipated. Participants will be included on the basis of physical examination, medical history, and vital signs performed between informed consent form (ICF) signature and vaccination
* Participant must be: a) postmenopausal (postmenopausal state is defined as no menses for 12 months without an alternative medical cause); and b) not intending to conceive by any methods
* Must sign an ICF indicating that the participant understands the purpose, procedures and potential risks and benefits of the study, and is willing to participate in the study
* Willing and able to adhere to the lifestyle restrictions specified in this protocol
* Agrees to not donate blood from the time of vaccination until 3 months after receiving the last dose of study vaccine

Exclusion Criteria:

* History of an underlying clinically significant acute or uncontrolled chronic medical condition or significant cognitive impairment or physical examination findings for which, in the opinion of the investigator, participation would not be in the best interest of the participant (for example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Known or suspected allergy or history of severe allergic reaction, anaphylaxis, or other serious adverse reactions to vaccines or vaccine excipients
* History of severe allergic reactions (for example anaphylaxis) to any component of the high-dose (HD) quadrivalent seasonal influenza vaccine, including egg protein, or following a previous dose of any influenza vaccine
* Has had major surgery (per the investigator's judgment) within 4 weeks before administration of the first study vaccine or will not have recovered from surgery per the investigator's judgment at time of vaccination
* History of acute polyneuropathy (for example, Guillain-Barré syndrome) or chronic inflammatory demyelinating polyneuropathy

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 959 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Hemagglutination Inhibition (HI) Antibody Titers Against Each of the Four Influenza Vaccine Strains as Measured by HI Assay | 29 days after High-dose (HD) quadrivalent influenza vaccination on Day 1 (Day 30)
  HI antibody titers measured by HI assay against each of the four influenza vaccine strains will be reported.
Antibody Titers to Vaccine O-serotype Antigens as Determined by Multiplex Electrochemiluminescent (ECL)-based Immunoassay 29 days After Administration of ExPEC9V on Day 1 | 29 days after administration of 9-valent extraintestinal pathogenic Escherichia coli vaccine (ExPEC9V) on Day 1 (Day 30)
  Antibody titers to vaccine O-serotype antigens as determined by multiplex ECL-based immunoassay 29 days after administration of ExPEC9V on Day 1 will be reported.
Antibody Titers to Vaccine O-serotype Antigens as Determined by Multiplex Electrochemiluminescent (ECL)-based Immunoassay 29 days After Administration of ExPEC9V on Day 30 | 29 days after administration of 9-valent extraintestinal pathogenic Escherichia coli vaccine (ExPEC9V) on Day 30 (Day 59)
  Antibody titers to vaccine O-serotype antigens as determined by multiplex ECL-based immunoassay 29 days after administration of ExPEC9V on Day 30 will be reported.

SECONDARY OUTCOMES:
Percentage of Seroconverted Participants | 29 days after HD quadrivalent influenza vaccination on Day 1 (Day 30)
  Percentage of seroconverted participants will be reported. Seroconversion is defined for each of the 4 influenza vaccine strains at 29 days after the administration of a HD quadrivalent seasonal influenza vaccine: 1) HI titer greater than or equal to (>=) 1:40 in participants with a pre-vaccination HI titer of less than (<) 1:10, or 2) a >=4-fold HI titer increase in participants with a pre-vaccination HI titer of >=1:10.
Percentage of Seroprotected Participants | 29 days after HD quadrivalent influenza vaccination on Day 1 (Day 30)
  Percentage of seroprotected participants will be reported. Seroprotection is defined for each of the 4 influenza vaccine strains as HI titer >=1:40 at 29 days after the administration of a HD quadrivalent seasonal influenza vaccine.
Percentage of Participants with Solicited Local (Injection Site) Adverse Events (AEs) for 14 Days After Each Vaccination | 14 days post-vaccination 1 on Day 1 (Day 15) and post-vaccination 2 on Day 30 (Day 44)
  Percentage of participants with solicited local (injection site) AEs for 14 Days after each vaccination will be reported. An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the study vaccination. Solicited local AEs are used to assess the reactogenicity of the study vaccine and are pre-defined local (injection site) and systemic events for which participants will be specifically questioned and which will be noted by participants in their participant diary for 14 days post vaccination (day of vaccination and the subsequent 14 days). Solicited local AEs are: injection site pain or tenderness, erythema and swelling at the study vaccine injection site. Solicited local AEs are considered related to study vaccine administration.
Percentage of Participants with Solicited Systemic AEs for 14 Days After Each Vaccination | 14 days post-vaccination 1 on Day 1 (Day 15) and post-vaccination 2 on Day 30 (Day 44)
  Percentage of participants with solicited systemic AEs for 14 Days after each vaccination will be reported. Solicited systemic AEs include following events: fatigue, headache, nausea, myalgia, and fever. Participants will be instructed on how to note signs and symptoms in the participant diary on a daily basis for 14 days post-vaccination (day of vaccination and the subsequent 14 days) for these events.
Percentage of Participants with Unsolicited AEs for 29 Days After Each Vaccination | 29 days post-vaccination 1 on Day 1 (Day 30) and post-vaccination 2 on Day 30 (Day 59)
  Percentage of participants with unsolicited AEs for 29 days after each vaccination will be reported. Unsolicited AEs are all AEs for which the participant is not specifically questioned in the participant diary.
Percentage of Participants with Medically-attended Adverse Events (MAAEs) From Vaccination 1 to Until 6 Months After Vaccination 2 | From vaccination 1 (on Day 1) till 6 months after vaccination 2 (on Day 30), that is until Day 210
  MAAEs are defined as AEs with medically-attended visits including hospital, emergency room, urgent care clinic, or other visits to or from medical personnel for any reason. AEs (for example, abnormal vitals) identified at a routine study visit will not be considered MAAEs.
Percentage of Participants with Serious Adverse Events (SAEs) From Vaccination 1 to Until 6 Months After Vaccination 2 | From vaccination 1 (on Day 1) till 6 months after vaccination 2 (on Day 30), that is until Day 210
  A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability or incapacity; congenital anomaly; is a suspected transmission of any infectious agent through a medicinal product; and is medically important.
Antibody Titers to Vaccine O-serotype Antigens and Exotoxin a Derived from Pseudomonas Aeruginosa (EPA) as Determined by Multiplex ECL-based Immunoassay | At days 1, 30, and 59
  Antibody titers to vaccine O-serotype antigens and EPA as determined by multiplex ECL-based immunoassay will be reported.
Opsonophagocytic Antibody Titers to Vaccine O-serotype Antigens as Determined by Multiplex Opsonophagocytic Assay (MOPA) 29 Days After Administration of ExPEC9V on Day 1 (Day 30) | 29 days after administration of ExPEC9V on Day 1 (Day 30)
  Opsonophagocytic antibody titers to vaccine O-serotype antigens as determined by MOPA 29 Days after administration of ExPEC9V on Day 1 (Day 30) will be reported.
Opsonophagocytic Antibody Titers to Vaccine O-serotype Antigens as Determined by Multiplex Opsonophagocytic Assay (MOPA) 29 Days After Administration of ExPEC9V on Day 30 (Day 59) | 29 days after administration of ExPEC9V on Day 30 (Day 59)
  Opsonophagocytic antibody titers to vaccine O-serotype antigens as determined by MOPA 29 Days after administration of ExPEC9V on Day 30 (Day 59) will be reported.
Antibody Titers to Vaccine O-serotype Antigens as Determined by Multiplex ECL-based Immunoassay 29 days after administration of ExPEC9V on Day 1 (Day 30) in participants with or without History of Urinary Tract Infection (UTI) at Enrollment | 29 days after administration of ExPEC9V on Day 1 (Day 30)
  Antibody titers to vaccine O-serotype antigens as determined by multiplex ECL-based Immunoassay will be reported 29 days after administration of ExPEC9V on Day 1 (Day 30) in participants with a history of UTI at enrollment and participants without a UTI history at enrollment
Antibody Titers to Vaccine O-serotype Antigens as Determined by Multiplex ECL-based Immunoassay 29 days after administration of ExPEC9V on Day 30 (Day 59) in participants with or without History of Urinary Tract Infection (UTI) at Enrollment | 29 days after administration of ExPEC9V on Day 30 (Day 59)
  Antibody titers to vaccine O-serotype antigens as determined by multiplex ECL-based Immunoassay will be reported 29 days after administration of ExPEC9V on Day 30 (Day 59) in participants with a history of UTI at enrollment and participants without a UTI history at enrollment
Opsonophagocytic Antibody Titers to Vaccine O-serotype Antigens as Determined by MOPA 29 days after administration of ExPEC9V on Day 1 (Day 30) in participants with or without History of UTI at Enrollment | 29 days after administration of ExPEC9V on Day 1 (Day 30)
  Opsonophagocytic antibody titers to vaccine O-serotype antigens as determined by MOPA 29 days after administration of ExPEC9V on Day 1 (Day 30) will be reported in participants with a history of UTI at enrollment and participants without a UTI history at enrollment.
Opsonophagocytic Antibody Titers to Vaccine O-serotype Antigens as Determined by MOPA 29 days after administration of ExPEC9V on Day 30 (Day 59) in participants with or without History of UTI at Enrollment | 29 days after administration of ExPEC9V on Day 30 (Day 59)
  Opsonophagocytic antibody titers to vaccine O-serotype antigens as determined by MOPA 29 days after administration of ExPEC9V on Day 30 (Day 59) will be reported in participants with a history of UTI at enrollment and participants without a UTI history at enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (41):
- United States (24):
  - Medical Affiliated Research Center Inc. (MARC), Huntsville, Alabama
  - Alliance for Multispeciality Research, Mobile, Alabama
  - Artemis Institute for Clinical Research, San Diego, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Optimal Research, Melbourne, Florida
  - Pharmax Research Clinic Inc, Miami, Florida
  - Suncoast Research Associates, LLC, Miami, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Velocity Clinical Research, Savannah, Georgia
  - Synexus Clinical Research US Inc, Chicago, Illinois
  - Optimal Research, Peoria, Illinois
  - Synexus Radiant Research, Inc, Evansville, Indiana
  - Heartland Research Associates, LLC, Newton, Kansas
  - Heartland Research Associates, an AMR Company, Wichita, Kansas
  - Alliance for Multispeciality Research, Lexington, Kentucky
  - Synexus Clinical Research US Inc, Creve Coeur, Missouri
  - Accellacare, Wilmington, North Carolina
  - CTI Clinical Trial and Consulting Services, Cincinnati, Ohio
  - Velocity Clinical Research, Cleveland, Ohio
  - Velocity Clinical Research, East Greenwich, Rhode Island
  - Alliance for Multispeciality Research, Knoxville, Tennessee
  - Benchmark Clinical Research - Austin, Austin, Texas
  - Optimal Research, Austin, Texas
  - Tekton Research Inc., Beaumont, Texas
- Belgium (3):
  - Universiteit Antwerpen - Centrum voor de Evaluatie van Vaccinaties (CEV), Edegem
  - Center for Vaccinology (CEVAC), Ghent
  - Az Sint-Maarten, Mechelen
- Canada (3):
  - Aggarwal and associates Ltd, Brampton, Ontario
  - Milestone Research, London, Ontario
  - Centricity Research- Manna Research (MR) - Quebec Location, Lévis, Quebec
- Poland (11):
  - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gdansk
  - PUNKT ZDROWIA Hlebowicz Jakubowski Lekarze sp.p., Gdansk
  - Synexus Polska Sp. z o.o. Oddzial w Gdynia, Gdynia
  - Synexus Polska Sp z o o Oddzial w Katowicach, Katowice
  - Pratia MCM Krakow, Krakow
  - Velocity Lublin, Lublin
  - Velocity Staszow, Staszów
  - MICS Centrum Medyczne Torun, Torun
  - MICS Centrum Medyczne Warszawa, Warsaw
  - Synexus Polska Sp z o o Oddzial w Warszawie, Warsaw
  - Synexus Polska Sp z o o Oddzial we Wroclawiu, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency